CLINICAL TRIAL: NCT01840072
Title: Inner Mongolia Stroke Project A Randomized Controlled Trial of Immediate Blood Pressure Reduction on Death and Major Disability in Patients With Acute Ischemic Stroke in China
Brief Title: China Antihypertensive Trial in Acute Ischemic Stroke
Acronym: CATIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Soochow University (Other)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Professor and Department Chair, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 140815
Record Dates: First submitted 2013-04-13; First posted 2013-04-25 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Hypertension; Antihypertensive Agents; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke; Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active antihypertensive treatment (Experimental): Active antihypertensive treatment
  Interventions: Other: Active antihypertensive treatment
- Usual care (No Intervention): Discontinue all home BP medications.

INTERVENTIONS:
Other: Active antihypertensive treatment — Initial antihypertensive treatment with angiotensin-converting enzyme inhibitors (Enalapril) and/or calcium channel blockers as second line medication; and/or diuretics as third line medications. Based on patients' baseline BP level, the first-line medication (intravenous Enalapril) can be used alone, or in combination with second-line medication (calcium channel blocker), and third-line medication (diuretics) to achieve the target systolic BP lowering by 10% to 25% within the first 24 hours after randomization and to achieve systolic BP below 140 mm Hg and diastolic BP below 90 mm Hg and maintain this BP level afterwards during the hospitalization.
  Arms: Active antihypertensive treatment

SUMMARY:
This randomized trial tests the effect of early blood pressure reduction on major disability and death among patients with acute ischemic stroke in china.

DETAILED DESCRIPTION:
We designed a randomized controlled clinical trial to test:

* The effectiveness of blood pressure reduction among patients with acute ischemic stroke (within 48 hours of onset) on the primary outcome, a combination of death within 14 days after randomization and dependency (modified Rankin scale ≥3) at 14 day or at the time of discharge, if that occurred before 14 days.
* The effectiveness of blood pressure reduction among patients with acute ischemic stroke (within 48-hours of onset) on secondary outcomes:

  * Combination of all-cause mortality and dependency over 3, 12, and 24 months of follow-up
  * Combined vascular disease events over 3, 12, and 24 months of follow-up (vascular deaths, non-fatal stroke, non-fatal myocardial infarction, coronary revascularization, hospitalized or treated angina, hospitalized or treated congestive heart failure, and hospitalized or treated peripheral arterial disease)
  * Recurrent fatal and non-fatal stroke over 3, 12, and 24 months of follow-up
  * Neurological functional status measured by NIH Stroke Score and modified Rankin scale at 14 day or discharge after randomization, and over 3, 12, and 24 months of follow-up
  * All-cause mortality over 3, 12, and 24 months of follow-up
  * Duration of initial hospitalization
  * Changes in systolic and diastolic blood pressure within 24 hours and over 7 days, and 14 days

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22 years
* Ischemic stroke onset within 48 hours confirmed by imaging (CT scan or MRI) study
* Systolic BP≥140 and <220 mm Hg and diastolic BP≥80 mm Hg
* No contraindications to antihypertensive treatment
* Able and willing to sign informed consent by patients or their direct family members

Exclusion Criteria:

* Individuals with hemorrhagic stroke
* Individuals with severe heart failure (NY Heart Association class III and IV), myocardial infarction, unstable angina, aortic dissection and cerebrovascular stenosis
* Individuals in a deep coma
* Individuals with resistant hypertension [systolic BP ≥170 mm Hg despite use of 4 or more antihypertensive medications for half a year or longer]
* Intravenous thrombolytic therapy (such as intravenous rtPA)
* Individuals who are unable to participate in follow-up examination
* Current pregnant women

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4071 (Actual)
Dates: Start 2009-08; Primary Completion 2013-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Principal Investigator — Tulane University SPHTM
Locations (1):
- Soohow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bu X, Li C, Zhang Y, Xu T, Wang D, Sun Y, Peng H, Xu T, Chen CS, Bazzano LA, Chen J, He J; CATIS Investigators. Early Blood Pressure Reduction in Acute Ischemic Stroke with Various Severities: A Subgroup Analysis of the CATIS Trial. Cerebrovasc Dis. 2016;42(3-4):186-95. doi: 10.1159/000444722. Epub 2016 Apr 26. PMID 27110711
- [Result] Zhong C, Xu T, Xu T, Peng Y, Wang A, Wang J, Peng H, Li Q, Geng D, Zhang D, Zhang Y, Zhang Y, Gao X, He J; CATIS Investigation Groups. Plasma Homocysteine and Prognosis of Acute Ischemic Stroke: a Gender-Specific Analysis From CATIS Randomized Clinical Trial. Mol Neurobiol. 2017 Apr;54(3):2022-2030. doi: 10.1007/s12035-016-9799-0. Epub 2016 Feb 24. PMID 26910818
- [Result] He J, Zhang Y, Xu T, Zhao Q, Wang D, Chen CS, Tong W, Liu C, Xu T, Ju Z, Peng Y, Peng H, Li Q, Geng D, Zhang J, Li D, Zhang F, Guo L, Sun Y, Wang X, Cui Y, Li Y, Ma D, Yang G, Gao Y, Yuan X, Bazzano LA, Chen J; CATIS Investigators. Effects of immediate blood pressure reduction on death and major disability in patients with acute ischemic stroke: the CATIS randomized clinical trial. JAMA. 2014 Feb 5;311(5):479-89. doi: 10.1001/jama.2013.282543. PMID 24240777
- [Result] Bu X, Zhang Y, Bazzano LA, Xu T, Guo L, Wang X, Zhang J, Cui Y, Li D, Zhang F, Ju Z, Xu T, Chen CS, Chen J, He J. Effects of early blood pressure reduction on cognitive function in patients with acute ischemic stroke. Int J Stroke. 2016 Dec;11(9):1009-1019. doi: 10.1177/1747493016660094. Epub 2016 Jul 13. PMID 27412188
- [Derived] Zhong C, Wang M, Liu D, Wei Y, Wang M, Peng Y, Chen J, Pan Y, Xu T, Wang Y, He J, Wang Y, Zhang Y, Liu L, Xie X. Antihypertensive Treatments After Acute Ischemic Stroke: to Continue or Not? Hypertension. 2026 Feb;83(2):e25575. doi: 10.1161/HYPERTENSIONAHA.125.25575. Epub 2025 Dec 5. PMID 41347304
- [Derived] Wang M, Long J, Yuan K, Cao M, Peng Y, Xu T, He J, Zhang Y, Zhong C, Zhai G. Soluble Triggering Receptor Expressed on Myeloid Cells 2 as a Promising Biomarker for Poststroke Depression After Acute Ischemic Stroke. J Am Heart Assoc. 2025 Sep 16;14(18):eJAHA2024040555T. doi: 10.1161/JAHA.124.040555. Epub 2025 Aug 22. PMID 40847526
- [Derived] Wang M, Zhu S, Long J, Cao M, Peng Y, Chen J, Xu T, He J, Zhang Y, Zhong C. Efficacy of immediate anti-hypertensive treatment in patients with acute ischaemic stroke stratified by mean arterial pressure and pulse pressure: a secondary analysis of the China Antihypertensive Trial in Acute Ischemic Stroke trial. Stroke Vasc Neurol. 2025 Dec 23;10(6):743-751. doi: 10.1136/svn-2024-003896. PMID 40268338
- [Derived] Wang Z, Zhang K, Zhong C, Zhu Z, Zheng X, Yang P, Che B, Lu Y, Zhang Y, Xu T. Plasma human cartilage glycoprotein-39 and depressive symptoms among acute ischemic stroke patients. Gen Hosp Psychiatry. 2025 May-Jun;94:120-125. doi: 10.1016/j.genhosppsych.2025.03.003. Epub 2025 Mar 6. PMID 40068363
- [Derived] Wang Z, Zhang K, Zhong C, Zhu Z, Zheng X, Yang P, Che B, Lu Y, Zhang Y, Xu T. Plasma Human Cartilage Glycoprotein-39 and Cognitive Impairment After Acute Ischemic Stroke. J Am Heart Assoc. 2025 Jan 21;14(2):e036790. doi: 10.1161/JAHA.124.036790. Epub 2025 Jan 17. PMID 39819010
- [Derived] He Y, Jia Y, Liu Y, Chang X, Yang P, Shi M, Guo D, Peng Y, Chen J, Wang A, Xu T, He J, Zhang Y, Zhu Z. High Plasma Polyamine Levels Are Associated With an Increased Risk of Poststroke Cognitive Impairment: A Multicenter Prospective Study From CATIS. J Am Heart Assoc. 2025 Jan 21;14(2):e037465. doi: 10.1161/JAHA.124.037465. Epub 2025 Jan 16. PMID 39817544
- [Derived] Sun L, Zhang Q, Shi M, Liu Y, Zhu Z, Zhang J, Peng H, Wang A, Chen J, Xu T, Zhang Y, He J. Associations Between Gene Variants of Lipid-Lowering Drug Targets and Adverse Outcomes After Ischemic Stroke. J Am Heart Assoc. 2024 Nov 19;13(22):e036544. doi: 10.1161/JAHA.124.036544. Epub 2024 Nov 15. PMID 39547981
- [Derived] Yang P, Shi M, Jia Y, Zhong C, Peng H, Sun L, Guo D, Chen J, Wang A, Xu T, Zhu Z, Zhang Y, He J. Plasma Polyamines and Short-Term Adverse Outcomes Among Patients With Ischemic Stroke: A Prospective Cohort Study. J Am Heart Assoc. 2024 Aug 6;13(15):e035837. doi: 10.1161/JAHA.124.035837. Epub 2024 Jul 31. PMID 39082415
- [Derived] Wang Z, Zhang K, Zhong C, Zhu Z, Zheng X, Yang P, Che B, Lu Y, Zhang Y, Xu T. Alcohol drinking modified the effect of plasma YKL-40 levels on stroke-specific mortality of acute ischemic stroke. Neuroscience. 2024 Aug 6;552:152-158. doi: 10.1016/j.neuroscience.2024.06.028. Epub 2024 Jun 27. PMID 38944147
- [Derived] Yang P, Wang S, Zhong C, Yin J, Yang J, Wang A, Xu T, Zhang Y. Association of Cardiac Biomarkers in Combination With Cognitive Impairment After Acute Ischemic Stroke. J Am Heart Assoc. 2024 Mar 5;13(5):e031010. doi: 10.1161/JAHA.123.031010. Epub 2024 Feb 23. PMID 38390800
- [Derived] Du J, Zhai Y, Dong W, Che B, Miao M, Peng Y, Ju Z, Xu T, He J, Zhang Y, Zhong C. One-Year Disability Trajectories and Long-Term Cardiovascular Events, Recurrent Stroke, and Mortality After Ischemic Stroke. J Am Heart Assoc. 2024 Feb 6;13(3):e030702. doi: 10.1161/JAHA.123.030702. Epub 2024 Jan 19. PMID 38240201
- [Derived] Zhai Y, Chen H, Che B, Liu Y, Peng Y, Chen J, Xu T, He J, Zhang Y, Zhong C. Efficacy of Immediate Antihypertensive Treatment in Patients With Acute Ischemic Stroke With Different Blood Pressure Genetic Variants. Hypertension. 2024 Mar;81(3):658-667. doi: 10.1161/HYPERTENSIONAHA.123.21851. Epub 2024 Jan 4. PMID 38174564
- [Derived] Zhai Y, Shi M, Liu Y, Peng Y, Zhu Z, Wang A, Peng H, Xu T, Chen J, Xu T, Zhang Y, He J, Zhong C. Magnitude of Systolic Blood Pressure Reduction and Early Achieved Blood Pressure and Clinical Outcomes After Acute Ischemic Stroke. J Am Heart Assoc. 2023 Oct 17;12(20):e030692. doi: 10.1161/JAHA.123.030692. Epub 2023 Oct 7. PMID 37804202
- [Derived] Zhu Z, Yang P, Jia Y, Wang Y, Shi M, Zhong C, Peng H, Sun L, Guo D, Xu Q, Chen J, Wang A, Xu T, He J, Zhang Y. Plasma Amino Acid Neurotransmitters and Ischemic Stroke Prognosis: A Multicenter Prospective Study. Am J Clin Nutr. 2023 Oct;118(4):754-762. doi: 10.1016/j.ajcnut.2023.06.014. Epub 2023 Aug 21. PMID 37793742
- [Derived] Zhu Z, Guo D, Zhang K, Yang P, Jia Y, Shi M, Peng Y, Chen J, Wang A, Xu T, Zhang Y, He J. Osteoprotegerin and Ischemic Stroke Prognosis: A Prospective Multicenter Study and Mendelian Randomization Analysis. Stroke. 2023 Feb;54(2):509-517. doi: 10.1161/STROKEAHA.122.040800. Epub 2022 Dec 13. PMID 36511149
- [Derived] Zhai Y, Che B, Liu Y, Peng H, Wang A, Peng Y, Chen J, Zhang Y, Xu T, Zhong C, He J. Effect of Immediate Antihypertensive Treatment on Clinical Outcomes in Acute Ischemic Stroke Patients With Different Renal Function Status. Hypertension. 2023 Jan;80(1):204-213. doi: 10.1161/HYPERTENSIONAHA.122.20202. Epub 2022 Nov 10. PMID 36353999
- [Derived] Du J, Miao M, Lu Z, Chen H, Bao A, Che B, Zhang J, Ju Z, Xu T, He J, Zhang Y, Zhong C. Plasma l-carnitine and risks of cardiovascular events and recurrent stroke after ischemic stroke: A nested case-control study. Nutr Metab Cardiovasc Dis. 2022 Nov;32(11):2579-2587. doi: 10.1016/j.numecd.2022.08.016. Epub 2022 Aug 28. PMID 36155150
- [Derived] Xu T, Zhang K, Zhong C, Zhu Z, Zheng X, Yang P, Che B, Lu Y, Zhang Y. Plasma Human Cartilage Glycoprotein-39 Is Associated With the Prognosis of Acute Ischemic Stroke. J Am Heart Assoc. 2022 Sep 20;11(18):e026263. doi: 10.1161/JAHA.122.026263. Epub 2022 Sep 14. PMID 36102255
- [Derived] Zang Y, Zhu Z, Shi M, Wang A, Xie X, Xu T, Peng Y, Yang P, Li Q, Ju Z, Geng D, Chen J, Liu L, Zhang Y, He J. Association between annual household income and adverse outcomes in patients who had ischaemic stroke. J Epidemiol Community Health. 2022 Mar;76(3):293-300. doi: 10.1136/jech-2021-216481. Epub 2021 Sep 7. PMID 34493532
- [Derived] Zhong C, Miao M, Che B, Du J, Wang A, Peng H, Bu X, Zhang J, Ju Z, Xu T, He J, Zhang Y. Plasma choline and betaine and risks of cardiovascular events and recurrent stroke after ischemic stroke. Am J Clin Nutr. 2021 Oct 4;114(4):1351-1359. doi: 10.1093/ajcn/nqab199. PMID 34159355
- [Derived] Che B, Shen S, Zhu Z, Wang A, Xu T, Peng Y, Li Q, Ju Z, Geng D, Chen J, He J, Zhang Y, Zhong C. Education Level and Long-term Mortality, Recurrent Stroke, and Cardiovascular Events in Patients With Ischemic Stroke. J Am Heart Assoc. 2020 Aug 18;9(16):e016671. doi: 10.1161/JAHA.120.016671. Epub 2020 Aug 11. PMID 32779506
- [Derived] Zhu S, Qian S, Xu T, Peng H, Dong R, Wang D, Yuan X, Guo L, Zhang Y, Geng D, Zhong C. White Matter Hyperintensity, Immediate Antihypertensive Treatment, and Functional Outcome After Acute Ischemic Stroke. Stroke. 2020 May;51(5):1608-1612. doi: 10.1161/STROKEAHA.119.028841. Epub 2020 Apr 1. PMID 32233741
- [Derived] Guo DX, Zhu ZB, Zhong CK, Bu XQ, Chen LH, Xu T, Guo LB, Zhang JT, Li D, Zhang JH, Ju Z, Chen CS, Chen J, Zhang YH, He J. Serum cystatin C levels are negatively correlated with post-stroke cognitive dysfunction. Neural Regen Res. 2020 May;15(5):922-928. doi: 10.4103/1673-5374.268928. PMID 31719258
- [Derived] Zhang R, Zhong C, Zhang Y, Xie X, Zhu Z, Wang A, Chen CS, Peng Y, Peng H, Li Q, Ju Z, Geng D, Chen J, Liu L, Wang Y, Xu T, He J. Immediate Antihypertensive Treatment for Patients With Acute Ischemic Stroke With or Without History of Hypertension: A Secondary Analysis of the CATIS Randomized Clinical Trial. JAMA Netw Open. 2019 Jul 3;2(7):e198103. doi: 10.1001/jamanetworkopen.2019.8103. PMID 31365109
- [Derived] Guo D, Zhu Z, Zhong C, Peng H, Wang A, Xu T, Peng Y, Xu T, Chen CS, Li Q, Ju Z, Geng D, Chen J, Zhang Y, He J. Increased Serum Netrin-1 Is Associated With Improved Prognosis of Ischemic Stroke. Stroke. 2019 Apr;50(4):845-852. doi: 10.1161/STROKEAHA.118.024631. PMID 30852966
- [Derived] He WJ, Zhong C, Xu T, Wang D, Sun Y, Bu X, Chen CS, Wang J, Ju Z, Li Q, Zhang J, Geng D, Zhang J, Li D, Li Y, Yuan X, Zhang Y, Kelly TN; CATIS investigators. Early antihypertensive treatment and clinical outcomes in acute ischemic stroke: subgroup analysis by baseline blood pressure. J Hypertens. 2018 Jun;36(6):1372-1381. doi: 10.1097/HJH.0000000000001690. PMID 29389742
- [Derived] Xu T, Zhang Y, Bu X, Wang D, Sun Y, Chen CS, Wang J, Peng H, Ju Z, Peng Y, Xu T, Li Q, Geng D, Zhang J, Li D, Zhang F, Guo L, Wang X, Cui Y, Li Y, Ma D, Zhang D, Yang G, Gao Y, Yuan X, Chen J, He J; CATIS investigators. Blood pressure reduction in acute ischemic stroke according to time to treatment: a subgroup analysis of the China Antihypertensive Trial in Acute Ischemic Stroke trial. J Hypertens. 2017 Jun;35(6):1244-1251. doi: 10.1097/HJH.0000000000001288. PMID 28169880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Antihypertensive Treatment | Usual Care
Started | 2038 | 2033
Completed | 2031 | 1986
Not Completed | 7 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Antihypertensive Treatment | Usual Care | Total
Number analyzed (Participants) | 2038 | 2033 | 4071
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.8) | 61.8 (11.0) | 62.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1317 | 1287 | 2604
  Male | 721 | 746 | 1467
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2038 | 2033 | 4071
Region of Enrollment [Number; unit: participants]
  China | 2038 | 2033 | 4071

OUTCOME MEASURES:

1. Primary Outcome: A Combination of Death Within 14 Days After Randomization and Major Disability at 14 Days or at Hospital Discharge if Earlier Than 14 Days.
Description: Major disability was defined as a score of 3 to 5 on the modified Rankin Scale at 14 days after randomization. Scores on the modified Rankin Scale range from 0 to 6, with a score of 0 indicating no symptoms; a score of 5 indicating severe disability (ie, bedridden, incontinent, or requiring constant nursing care and attention); and a score of 6 indicating death.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Usual Care | Active Antihypertensive Treatment
Number analyzed (Participants) | 2033 | 2038
participants | 681 | 683

2. Secondary Outcome: A Combination of All-cause Mortality and Major Disability at the 3-month Post-treatment Follow-up.
Description: Major disability was defined as a score of 3 to 5 on the modified Rankin Scale at 3 months after randomization. Scores on the modified Rankin Scale range from 0 to 6, with a score of 0 indicating no symptoms; a score of 5 indicating severe disability (ie, bedridden, incontinent, or requiring constant nursing care and attention); and a score of 6 indicating death
Time Frame: 3 months
Population: All participants examined at 3-month posttreatment follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Active Antihypertensive Treatment
Number analyzed (Participants) | 1987 | 1988
Participants | 502 | 500

3. Secondary Outcome: Mortality
Description: Those patients who are still alive at hospital discharge will be contacted by telephone to set up a follow-up clinical visit. Information on clinical deaths will be obtained.
Time Frame: 3 months
Population: All participants followed at 3-month posttreatment follow-up visit
Measure: Number; unit: participants
Arm/Group | Active Antihypertensive Treatment | Usual Care
Number analyzed (Participants) | 1988 | 1987
participants | 68 | 54

4. Secondary Outcome: Recurrent Stroke
Description: Those patients who are still alive at hospital discharge will be contacted by telephone to set up a follow-up clinical visit. Information of recurrent stroke will be collected.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Active Antihypertensive Treatment | Usual Care
Number analyzed (Participants) | 1988 | 1987
participants | 28 | 43

5. Secondary Outcome: Other Vascular Events
Description: Those patients who are still alive at hospital discharge will be contacted by telephone to set up a follow-up clinical visit. Information of vascular events, such as myocardial infarction, will be collected.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Usual Care | Active Antihypertensive Treatment
Number analyzed (Participants) | 1987 | 1988
participants | 59 | 48

6. Secondary Outcome: Long-term Neurological and Functional Status
Description: Those patients who were still alive at hospital discharge were contacted by telephone to set up a follow-up clinical visit. Neurological function was assessed by the modified Rankin scale at the 3-month post-treatment follow-up visit. Scores on the modified Rankin Scale range from 0 to 6, with a score of 0 indicating no symptoms; a score of 5 indicating severe disability (ie, bedridden, incontinent, or requiring constant nursing care and attention); and a score of 6 indicating death. Major disability was defined as a score of 3 to 5 on the modified Rankin Scale.
Time Frame: Three months
Population: Those patients who are still alive and followed at 3-Month posttreatment follow-up visit
Measure: Median (Inter-Quartile Range); unit: Score on modified Rankin scale
Arm/Group | Usual Care | Active Antihypertensive Treatment
Number analyzed (Participants) | 1987 | 1988
Score on modified Rankin scale | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]

7. Secondary Outcome: Cognitive Function (the Mini-Mental State Examination)
Description: Cognitive function was measured by the Mini-Mental State Examination at 3 months after randomization. The MMSE contains 20 items that test cognitive performance in domains including orientation, registration, attention and calculation, recall, language, and visual construction. MMSE scores were divided into three ordinal categories: 24-30 (no cognitive impairment), 19-23 (mild cognitive impairment), and 0-17 (severe cognitive impairment).
Time Frame: Three months
Population: In a pre-planned ancillary study, 660 participants were systemically selected prior to randomization for cognitive function assessment. At the 3-month visit, 15 patients were lost to follow-up and 7 patients were deceased. A total of 638 participants who completed the cognitive function tests were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: MMSE score
Arm/Group | Usual Care | Active Antihypertensive Treatment
Number analyzed (Participants) | 324 | 314
MMSE score | 26 [22 to 29] | 26 [22 to 29]

8. Secondary Outcome: Cognitive Function (Montreal Cognitive Assessment)
Description: Cognitive function was measured by Montreal Cognitive Assessment at 3 months after randomization. The MoCA is a 30-item test that evaluates the following seven cognitive domains: visuospatial/executive functions, naming, memory, attention, language, abstraction, and orientation. One point is added for participants with education <12 years. Scores on the MoCA range from 0 to 30 and cognitive impairment was defined as a score of <26.
Time Frame: Three months
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: MoCA score
Arm/Group | Usual Care | Active Antihypertensive Treatment
Number analyzed (Participants) | 324 | 314
MoCA score | 22 [18 to 26] | 22 [18 to 26]

9. Secondary Outcome: Quality of Life
Description: Due to limited funding, quality of life data were not collected.
Time Frame: 3 months
Arm/Group | Usual Care | Active Antihypertensive Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days, 3 months, 12 months, and 24 months
Description: No serious or other (non-serious) adverse events were observed for any participants.
Arm/Group | Active Antihypertensive Treatment | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/2038 | 0/2033
Other Adverse Events (participants affected / at risk) | 0/2038 | 0/2033

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes